CLINICAL TRIAL: NCT01843712
Title: Study of Eating in the Absence of Hunger and of Caloric Compensation in French Children, and of Their Relationships With Parental Feeding Practices
Brief Title: Eating in the Absence of Hunger and Caloric Compensation in Preschool Children, Link With Parental Feeding Practices
Acronym: HabEatWP31
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: HabeatWP31; WP31.INRA (Other: INRA)
Record Dates: First submitted 2013-04-16; First posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Food Intake Regulation in Healthy Children
Keywords: Caloric compensation; Eating in the absence of hunger; Children; Parental feeding practices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objectives: The aims were to measure caloric compensation (CC) and eating in the absence of hunger (EAH) in 2 to 7 year-old French children in their regular eating context and to link these measurements with individual characteristics (adiposity, age, gender) and parental feeding practices.

Design: Three consecutive weeks an identical lunch was served in four preschool canteens reaching 236 children. The first lunch was a control session. For the CC situation (week 2), thirty minutes before the lunch children were offered a preload (137 kcal). For the EAH situation (week 3), ten minutes after lunch children were exposed to palatable foods (430 kcal). Food intake was measured at the individual level. Parental eating behaviour and feeding practices were measured by questionnaires. Child's height and weight were measured by a medical doctor.

ELIGIBILITY:
Inclusion Criteria:

* To be registered to the school canteen, to provide parental approval

Exclusion Criteria:

* Chronic disease or food allergies.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population was composed of 236 children aged 2 to 7 years-old
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Caloric compensation measurement | 1 week
  In order to collect measurements of caloric compensation, children were offered a chocolate bun 30 minutes before the lunch on the second week. The food intake at lunch was recorded. We calculated if children compensated the chocolate bun, by comparing energy intake at this lunch with energy intake from the control lunch which took place on week 1.
Control measurement of energy intake | 1 week
  The first week, we conducted a control lunch and recorded food intake of each child.
Eating in the absence of hunger measurement | 1 week
  In order to collect the measurement of Eating in the absence of hunger, on the third week we offered palatable foods to children 10 minutes after their lunch. We recorded the energy intake from these post-meal foods.

SECONDARY OUTCOMES:
Parental feeding practices | One month after inclusion
  Using a validated questionnaire, we collected information about parental feeding practices (Comprehensive Feeding Practices Questionnaire, Musher-Eizenman & Holub, 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Nicklaus Sophie, phD, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Centre des sciences du goût et de l'alimentation, Dijon, France

REFERENCES:
- [Derived] Remy E, Issanchou S, Chabanet C, Boggio V, Nicklaus S. Impact of adiposity, age, sex and maternal feeding practices on eating in the absence of hunger and caloric compensation in preschool children. Int J Obes (Lond). 2015 Jun;39(6):925-30. doi: 10.1038/ijo.2015.30. Epub 2015 Mar 17. PMID 25777357
- See also: Web site for the main research project funded by the European Union — http://www.habeat.eu/